CLINICAL TRIAL: NCT05045677
Title: Digital Dialectical Behavioral Therapy (d-DBT) Skills for Treatment of Acute Suicidality in Psychiatric Inpatients: Randomized Feasibility Trial
Brief Title: Digital Dialectical Behavioral Therapy (d-DBT) Skills for Acute Suicidality in Psychiatric Inpatients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 047-2021
Record Dates: First submitted 2021-08-09; First posted 2021-09-16 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Suicidal Ideation
MeSH Terms: conditions — Suicidal Ideation | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital DBT intervention group (Experimental): Digital intervention group plus standard care
  Interventions: Other: digital DBT skills intervention; Other: Standard Care
- Standard care (Active Comparator): Standard care alone
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: digital DBT skills intervention — The digital intervention consists of 6 modules that will be delivered over 6 to 10 days. The modules cover mindfulness skills, emotion regulation skills and distress tolerance skills.
  Arms: Digital DBT intervention group
Other: Standard Care — Standard inpatient care includes a multi-disciplinary team approach including daily psychiatric review, medication management and in-person psychosocial interventions (social work, nursing).

SUMMARY:
Suicidality (ideation about taking one's life, suicide plans, and attempts) is a major public health concern in Ontario and worldwide. Psychiatric inpatients with suicidality represent a group that is high-risk for subsequent suicide. Current standard-care for suicidal psychiatric inpatients focuses on containment of risk and indirect treatment of suicidality by treating any underlying mental disorder. Though there is evidence that addressing suicidality directly is more effective than an indirect approach, there are limited evidence based treatments that target suicidality. Furthermore, there are few high-quality studies that have included inpatients. Psychotherapeutic interventions are under-utilized for inpatients and COVID-19 has further widened this gap given attempts by hospitals to reduce face-to-face contact with patients. Digital psychotherapy interventions have the ability to bridge this gap given their lower cost, ease of dissemination, acceptability by patients, and effectiveness. To our knowledge, there are no studies that have assessed the feasibility, acceptability and effectiveness of digital interventions for suicidal inpatients. Our study is a feasibility trial of a previously studied digital Dialectical Behavioural Therapy (d-DBT) skills intervention in suicidal psychiatric inpatients.

The study is a two arm randomized parallel group-controlled trial, 6-10 day, flexible timeline, randomized feasibility trial of a d-DBT skills intervention added to standard care for patients admitted to psychiatric inpatient units with suicidality. There will be 20 patients who will receive the intervention in addition to standard care and 20 patients who will receive standard care alone. There will also be a 4 week follow-up after discharge from hospital.

Participants will be admitted for psychiatric care at the Complex and Critical Care Units, Centre for Addiction and Mental Health (CAMH), Toronto.

ELIGIBILITY:
Inclusion Criteria:

1. patients with any DSM-5 diagnosis aged 18 years and above;
2. admitted to CAMH with suicidality and a baseline BSI score of > 6;
3. capable and willing to give informed consent;
4. anticipated length of admission is greater than 5 days;
5. deemed suitable by the primary team to take part in a psychotherapeutic intervention as part of standard care

Capacity to consent will be evaluated by the research staff performing the informed consent process. It will be assessed as the participant's ability to understand and appreciate the risks and benefits of taking part in the proposed study.

Exclusion Criteria:

1. presence of psychiatric symptoms that interfere with the ability to complete the d-DBT
2. Concurrent treatment with ECT or MST

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Recruitment and retention rates | 6-10 days
  Feasibility - whether the intervention is possible in the acute inpatient setting
Client Satisfaction Questionnaire 8 (CSQ-8) | 6-10 days
  Acceptability - whether the intervention is appropriate for the acute inpatient setting. The CSQ-8 scores range from 8 to 32, with higher values indicating higher satisfaction with the intervention.
User Experience Questionnaire (UXQ) | 6-10 days
  Usability - whether the intervention is serviceable for its intended purpose. The UXQ has 11 items exploring characteristics informing usability of mobile apps, each scored from 0-10, for a total score ranging from 10-110 (with larger scores indicating increased usability).

SECONDARY OUTCOMES:
Columbia-Suicide Severity Rating Scale (C-SSRS) | 5-10 days in addition to discharge and 4 weeks post-discharge
  Preliminary efficacy - whether symptoms of suicidal ideation are reduced by the intervention. The sum ranges from 2 to 25, with the higher number indicating more intense ideation.
Clinical Global Impression (CGI) | 5-10 days in addition to discharge and 4 weeks post-discharge
  Preliminary efficacy - whether CGI change during the clinical trial. The CGI asks the clinician to rank the current severity of illness and global improvement. Scores range form 1 to 7 with a higher score corresponding to more severe illness
Brief Difficulties in Emotion Regulation Scale (DERS-16) | 5-10 days in addition to discharge and 4 weeks post-discharge
  Preliminary efficacy - whether symptoms of emotion regulation change during the trial. Total scores on the DERS-16 can range from 16 to 80, with higher scores reflecting greater levels of emotion dysregulation
Kessler psychological distress scale (K10) | 5-10 days in addition to discharge and 4 weeks post-discharge
  Preliminary efficacy - whether symptoms of distress are improved by the intervention. Scores range from 10 to 50, with increasing scores indicating increasing distress and severity of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Ishrat Husain, MD (Res), Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No